CLINICAL TRIAL: NCT03652480
Title: Efficacy and Safety of Subacromial Corticosteroid Injection in Type-2 Diabetic
Brief Title: Shoulder Corticosteroid Injection in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Enrico Bellato, Researcher, University of Turin, Italy
Other Study IDs: SHOULDERDM2013
Record Dates: First submitted 2018-08-25; First posted 2018-08-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Shoulder Pain; Corticosteroid Injection; Type2 Diabetes Mellitus
Keywords: shoulder pain; type 2 diabetes; subacromial corticosteroid injection; glycemia; efficacy; safety
MeSH Terms: conditions — Shoulder Pain; Diabetes Mellitus, Type 2 | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: MethylPREDNISolone Acetate 40 MG/ML

SUMMARY:
In type 2 diabetic patients affected by chronic shoulder pain, subacromial injection with corticosteroid could be an effective treatment. The aim of this study was to measure the risk-benefit ratio of this treatment.Twenty patients with well-controlled diabetes were included in a prospective study. In a first pre-injection phase, patients were asked to measure glycemia for 7 days, before breakfast and dinner, then 2 hours after lunch and dinner. Baseline data including Constant Score (CS), Subjective Shoulder Value (SSV) and Numerical Rating Scale (NRS) for pain were collected. Patients were treated with subacromial injection with 40mg of Methylprednisolone Acetate and 2ml of Lidocaine. At discharge, patients were asked to re-measured glycemia for the following week.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study.
* Severe overall pain and night pain: Numerical Rating Scale (NRS) for pain[8] above or equal to 60/100; the scale was modified from 0-10 to 0-100 (0 = no pain 100 = unbearable pain).
* No significant improvement after at least 2 courses of physiotherapy (including direct assistance from a physical therapist with specific exercises, manual therapy, and physical agents in order to reduce inflammation and pain).
* Clinical signs of subacromial tendinobursitis, with or without signs of rotator cuff tear, defined as positive Neer, Yocum and Hawkins tests[9-15]. Pain experienced during the execution of these tests needed to reproduce the type of pain that patients complained the most.
* No indication for surgery due to the age, concomitant comorbidities or patient's refusal to undergo surgery.
* Well-controlled type-2 diabetes, defined as:

  * Fasting and pre-prandial blood glucose levels in the range of 90- 150mg/dL.
  * Hb1Ac <64mmol/mol (corresponding to 8%) measured within 6 months.
* A device for self-measurement of blood sugar levels at home
* Patients need to have a recent (within 6 months) x-ray and an MRI or ultrasound of the affected shoulder

Exclusion Criteria:

* Corticosteroid treatment in the past 3 months.
* Complaints of shoulder stiffness more than shoulder pain.
* Symptomatic glenohumeral arthritis defined as shoulder stiffness plus moderate radiographic signs of arthritis (grade >2 according to Hamada classification and grade >1 according to Samilson-Prieto classification for eccentric and concentric arthritis respectively).
* Shoulder trauma within 3 months of inclusion evaluation for in this study.
* High blood pressure values (systolic blood pressure >140mmHg, diastolic blood pressure >80mmHg).
* Glaucoma.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type-2 diabetic patients affected complaining of chronic shoulder pain resistant to at least 6 months of conservative therapy (NSAIDs, painkillers and physiotherapy).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemia | Patients were requested to measure their blood sugar levels 4 times a day for the following 7 days
  Post-injections glucose blood levels (mg/dl)

SECONDARY OUTCOMES:
Constant Score (CS) | 30 days post-injection, 6 months post-injection
  The CS is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.
  Subjective findings (severity of pain, activities of daily living and working in different positions) of the participants are responsible for 35 points and objective measurements (active range of motion without pain, measurements exo -and endorotation via reference points and measuring muscle strength) are responsible for the remaining 65 points.
Oxford Shoulder Score (OSS) | 30 days post-injection, 6 months post-injection
  The OSS questionnaire contains 12 items, each with five potential answers. Patients are asked to rate their symptoms between 1 (minimal symptoms) and 5 (severe symptoms). The combined total gives a minimum score of 12 and a maximum of 60
Subjective Shoulder Value (SSV) | 30 days post-injection, 6 months post-injection
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%
Subjective Outcomes Determination (SOD) score | 30 days post-injection, 6 months post-injection
  The SOD score is a simple tool with a categorical and a numerical component to compare surgical outcomes to both the preoperative status as well as to the preinjury state. Patients are asked to compare how they feel currently to how they felt before their surgery and to state if they overall consider themselves to be better, worse ore they are not sure. If they feel better, they are asked to indicate if they consider the operated part of the body to be Improved, Greatly improved, Almost Normal, or Normal. If they feel worse, the respondent is asked if they are Worse, Profoundly Worse, or As Bad As Dying

REFERENCES:
- [Derived] Blonna D, Bonasia DE, Mattei L, Bellato E, Greco V, Rossi R. Efficacy and Safety of Subacromial Corticosteroid Injection in Type 2 Diabetic Patients. Pain Res Treat. 2018 Sep 20;2018:9279343. doi: 10.1155/2018/9279343. eCollection 2018. PMID 30327731